CLINICAL TRIAL: NCT03993990
Title: Effects of Empowerment-based Program on Post-discharge Self-care Behavior, Glycemic Control, and Prevention of Foot Ulcer Infection and Occurrence in Patients With Diabetic Foot Ulcer
Brief Title: Effects of Empowerment-based Program on Post-discharge Glycemic Control, and Foot Ulcer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial resources
Sponsor: Chin yenfan (Other)
Responsible Party: Sponsor-Investigator, Chin yenfan, assistant professor, Chang Gung Memorial Hospital
Organization: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201802180B0
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetes、Foot ulcer、Self-care、glycemic control、Empowerment
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants will receive an empowerment-based intervention individually, based on five steps (i. e. problem identification, meaning and perception clarification, intervention planning, intervention delivery, and evaluation).
  Interventions: Behavioral: individual empowerment-based intervention
- Control group (No Intervention): Participants will receive routine care of the research setting only. The counseling will be provided if participants request.

INTERVENTIONS:
Behavioral: individual empowerment-based intervention — Participants will receive an empowerment-based intervention individually, based on five steps (i. e. problem identification, meaning and perception clarification, intervention planning, intervention delivery, and evaluation). After the principal investigator delivers a pre-discharge assessment (i. e. the self-care behavior and self-efficacy of diabetes and diabetic foot ulcer, risk factors of foot ulcer, family support, and threat belief of participant), the plan of behavioral modification will be determined by the principal investigator and participants. The subsequent follow-up and intensifying interventions will be delivered at the following time points: three days after discharge, every weeks for one month, every two weeks for subsequent two months, and then every three months for three times.
  Arms: Experimental group

SUMMARY:
The purpose of this study is to evaluate an empowerment-based program. A randomized controlled trial design will be used. From August 2019 to July 2021, 160 subjects will be recruited at a medical center and randomly assigned to the intervention or comparison group. Participants in the intervention group will receive an assessment of their self-care demand and self-efficacy, as well as an empowerment-based program delivered by the project host. The program includes the identification of the problems of participants, clarification of their feelings and the significance of their problems, plan setting discussion, motivation for action, and evaluation of the execution of their plan. Empowerment-based strategies will be provided individually at the following time points: before discharge, on post-discharge days 3, 7, 14, 21, 28, 42, 56, 70, and 84, and at 6, 9, and 12 months post-discharge. Those in the comparison group will receive routine care only. Outcome measures include self-care behaviors, glycemic control (measured by HbA1C), diabetic foot ulcer infection, and diabetic foot ulcer recurrence. Data will be collected at baseline and at 1, 3, 6, and 12 months after discharge.

DETAILED DESCRIPTION:
A randomized controlled trial design will be used to evaluate an empowerment-based program.. From August 2019 to July 2021, 160 subjects will be recruited at a medical center and randomly assigned to the intervention or comparison group. Participants in the intervention group will receive an assessment of their self-care demand and self-efficacy, as well as an empowerment-based program delivered by the project host. The program includes the identification of the problems of participants, clarification of their feelings and the significance of their problems, plan setting discussion, motivation for action, and evaluation of the execution of their plan. Empowerment-based strategies will be provided individually at the following time points: before discharge, on post-discharge days 3, 7, 14, 21, 28, 42, 56, 70, and 84, and at 6, 9, and 12 months post-discharge. Those in the comparison group will receive routine care only. Outcome measures include self-care behaviors, glycemic control (measured by HbA1C), diabetic foot ulcer infection, and diabetic foot ulcer recurrence. Data will be collected at baseline and at 1, 3, 6, and 12 months after discharge

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Age between 20 and 80 years old.
* Could communicate with Mandarin or Taiwanese.
* The glycated hemoglobin value is higher or equal to 7.5%.
* The vibration or monofilament test results are abnormal.
* Wagner stage 1 or 2 foot ulcer
* The location of ulcer is at the big toes or on the sole

Exclusion Criteria:

* Cognitive impairment
* Severe lower extremity arterial insufficiency disease
* Osteomyelitis or foot ulcer recurrent
* Alcoholism or Drug addiction
* Autoimmune disease
* Unable to perform daily self-care activity
* The main caregivers are foreigner and no other family members live together
* The C-reactive protein values are higher than 15 mg/dL
* Admitting in a long-term care institution after discharge from hospital
* No intention of the return-visit at the clinic of research hospital

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | Less than 1 minute
  Glycated hemoglobin value
Foot infection and recurrence of foot ulcer | 5 minutes
  Foot assessment and the review of medical record

SECONDARY OUTCOMES:
Knowledge regarding warning signs of diabetic foot ulcer | 5 minutes
  The WS-DFUD-KQ comprises of 12 items. Three of the 12 items are negatively worded and state as misconceptions regarding warning signs of diabetic foot ulcer deterioration (i.e. item 8, 9, 10). The response choices include "yes," "no," and "uncertain." Each item with the correct answer obtains a score of 1, after which the scores are summed to obtain a total score.
Self-care behaviors of foot care | 3 minutes
  The Diabetes Foot Self-Care Behavior Scale (DFSBS) The DFSBS contains 7 items. The scale had two parts: In the first part, the responses were rated on the number of days patients performed a certain behavior over the course of one week. In the second part, the responses were rated by the frequency with which patients performed a certain behavior in general, from never (1) to always (5).
Self-care behaviors of diabetes | 4 minutes
  The Chinese version of summary of diabetes self-care activity questionnaire (C-SDSCA) The C-SDSCA is a short self-reported questionnaire of diabetes self-management across five components of diabetes regimen a person with diabetes should practice in order to stay well ( i. e. diet, exercise, blood sugar testing, foot care and attention to smoking.)
Diabetes-related Foot Ulcer Self-Management Behavior | 9 minutes
  The Diabetes-related Foot Ulcer Self-Management Behavior Scale (DFUSMBS) measures behaviors that patients use to manage their diabetes-related foot ulcers to promote wound healing and to prevent the deterioration of their wounds, including timely treatment seeking and management, wound management, and self-management of diabetes. The 18-item scale includes three reverse-scored items (Item 1, 2, 11) and uses a 5-point Likert scale (1 = never, 2 = seldom, 3 = sometimes, 4 = frequently, and 5 = always).
Diabetes Management Self-Efficacy | 10 minutes
  The Chinese version of the Diabetes Management Self-Efficacy Scale (C-DMSES) was a self-administered scale containing 20 items. It assessed the extent to which respondents were confident that they could manage their blood sugar, diet, and level of exercise. Responses were rated on a 10-point Likert-style from not at all (1) to certainly can do (10). The responses were summed to become a total score for "self-efficacy". Possible scores ranged from 0 to 200 points. The tool had acceptable reliability and validity in a Taiwanese population.
Self-efficacy regarding diabetes foot self-car | 1 minutes
  Two items were used to measure the self-efficacy regarding diabetes foot self-care of participants. They are "I have confidence to check my feet (including the bottom of my feet and between the toes) daily, either by myself or to ask for someone's help.", and "I have confidence to apply moisturizing lotion to my feet by myself or asking for someone's help, If my skin is dry". Responses were rated on a 10-point Likert-style scale according the degree of confidence.
Self-efficacy regarding diabetes-related foot ulcer self-management | 5 minutes
  The 16-item diabetes-related foot ulcer self-management self-efficacy scale was used to measure the confidence in delivering diabetic foot ulcer self-management behavior, and management of diabetic foot ulcer. Responses were rated on a 10-point Likert-style from not at all (1) to certainly can do (10). The higher score indicates better self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Yenfan Chin, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No